CLINICAL TRIAL: NCT03406715
Title: Combination Immunotherapy With Ipilimumab and Nivolumab Plus a Dendritic Cell Based p53 Vaccine (Ad.p53-DC) in Patients With Relapsed Small Cell Lung Cancer (SCLC)
Brief Title: Combination Immunotherapy-Ipilimumab-Nivolumab-Dendritic Cell p53 Vac - Patients With Small Cell Lung Cancer (SCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor closed study
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry); MultiVir, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19163; CA209-9KN (Other: Bristol-Myers Squibb Protocol Number); MVIR-Adp53DC-001 (Other: MultiVir, Inc. Protocol Number)
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Results first posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Small Cell Lung Cancer; Lung Cancer; Relapsed Small Cell Lung Cancer
Keywords: SCLC; Lung Cancer; Lung Disease; Relapsed SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms; Lung Diseases | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Immunotherapy Plus Vaccine (Experimental): Combination immunotherapy with Ipilimumab and Nivolumab plus a Dendritic Cell based p53 Vaccine (Ad.p53-DC). Induction Immunotherapy, followed by Maintenance Immunotherapy and potentially Retreatment. During retreatment, participants would receive the combination of Ipilimumab and Nivolumab or Nivolumab alone every three weeks for a maximum of one additional year.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Biological: Dendritic Cell based p53 Vaccine

INTERVENTIONS:
Drug: Nivolumab — Nivolumab (BMS-936558) is an anti-PD-1 antibody. It works by attaching to and blocking a molecule called PD-1. Induction Immunotherapy Phase (4 x 21 days cycles): Nivolumab on Day 1 of each cycle for 4 cycles. Maintenance Immunotherapy beginning on Day 1 of Cycle 5: Nivolumab only on Day 1 of every 4 week period. Participants will continue to receive Nivolumab only on Day 1 of each additional 4 week period that they take part until their disease progresses. The Retreatment phase of the study may be available to participants whose doctor feels they would benefit from retreatment and if they qualify for this retreatment.
  Other Names: BMS-936558
Drug: Ipilimumab — Ipilimumab is an antibody (a type of human protein) that is approved to treat patients with metastatic melanoma. In this study, the use of ipilimumab is investigational. Induction Immunotherapy Phase (4 x 21 days cycles): Ipilimumab on Day 1 of each cycle for 4 cycles. The Retreatment phase of the study may be available to participants whose doctor feels they would benefit from retreatment and if they qualify for this retreatment.
  Other Names: Yervoy®
Biological: Dendritic Cell based p53 Vaccine — Dendritic Cell based p53 Vaccine (Ad.p53-DC). The p53 vaccine will be made by inserting the p53 gene (a gene is a hereditary unit of all living organism within a cell) into a subset of the participant's own white blood cells. The insertion of the gene into their white blood cells will occur in the laboratory, after their cells have been extracted from their body through a procedure called leukopheresis (similar to dialysis). Induction Immunotherapy Phase (4 x 21 day cycles): Participants will receive the p53 vaccine on Days 1 and 15 of cycle 1 and then again on Day 8 of Cycle 2. Maintenance Immunotherapy beginning on Day 1 of Cycle 5: p53 vaccine three additional times (every 4 weeks over a 12 week period).
  Other Names: Ad.p53-DC

SUMMARY:
The purpose of this study is to find out what effects (good and bad) immunotherapy treatment using the p53 vaccine (Ad.p53-DC) in combination with Nivolumab and Ipilimumab has on small cell lung cancer. Immunotherapy is a cancer therapy that uses the body's immune system to fight cancer cells.

This study can be divided into three different phases: initial Induction Immunotherapy, Maintenance Immunotherapy and Retreatment.

DETAILED DESCRIPTION:
During the Induction Immunotherapy phase (4 x 21 day cycles) of the study, participants will receive Ipilimumab and Nivolumab on Day 1 of each cycle for 4 cycles. Participants will receive the p53 vaccine on Days 1 and 15 of cycle 1 and then again on Day 8 of Cycle 2.

Beginning on Day 1 of Cycle 5 participants will start Maintenance Immunotherapy. During this phase of the study, participants will receive Nivolumab only on Day 1 of every 4 week period. Participants will also receive the p53 vaccine three additional times (every 4 weeks over a 12 week period). During Maintenance Immunotherapy you will continue to receive Nivolumab only on Day 1 of each additional 4 week period that you take part until your disease progresses.

The Retreatment phase of the study may be available to participants whose doctor feels they would benefit from retreatment and if they qualify for this retreatment. During retreatment, participants would receive the combination of Ipilimumab and Nivolumab or Nivolumab alone every three weeks for a maximum of one additional year.

P53 Vaccine production

The p53 vaccine will be made by inserting the p53 gene (a gene is a hereditary unit of all living organism within a cell) into a subset of the participant's own white blood cells. The insertion of the gene into their white blood cells will occur in the laboratory, after their cells have been extracted from their body through a procedure called leukopheresis (similar to dialysis).

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of SCLC
* Recurrence to at least one prior treatment with a platinum containing regimen (cisplatin or carboplatin) including limited stage (LS) and extensive stage (ES) initial presentations. Note: In patients with SCLC the most frequent platinum containing doublet used is etoposide-carboplatin. However, etoposide-cisplatin and irinotecan or topotecan combined with either carboplatin or cisplatin are platinum doublet regimens that can sometimes be used and thus would be allowed for the purposes of trial enrollment and eligibility.
* Excluded are patients who upon relapse may be still considered for a salvage concurrent chemo-radiation approach.
* Willing and able to provide written informed consent/assent for the trial.
* Be 18 years of age or older on day of signing informed consent
* Have measurable disease based on Response Evaluation in Solid Tumors (RECIST) 1.1
* Have a performance status of 0 - 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Demonstrate adequate organ function. All screening labs should be performed within 30 days of treatment initiation.
* Life expectancy of >4 months.
* Favorable tumor p53 biomarker profile defined by ≥ 50% p53 positive tumor cells by immunohistochemistry. Tumor p53 biomarker evaluations may be performed with either original or recurrent tumor although samples from recurrent disease are preferred.
* Females of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Females of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication.
* Males should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Therapy: Systemic steroid doses of less than 10 mg of prednisone daily or its equivalent are allowed in patients receiving physiologic replacement steroid doses for both criteria 2 and 8.
* Has a known history of active Bacillus Tuberculosis (TB)
* Hypersensitivity to Ipilimumab and/or nivolumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) excluding any anti-PD-1 and/or anti-PD-L1 checkpoint inhibitor within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. - Note: Potential participants with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. - Note: If potential participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer. Other malignancies that remain without evidence of disease or recurrence, 2 years or more after curative therapy are also considered part of this exception.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 2 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Any diagnosis of autoimmune disease (confirmed by medical records or appropriate laboratory testing)
* Known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with participation for the full duration of the trial, or is not in the best interest of the person to participate, in the opinion of the treating investigator.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
* Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Excluded are patients who upon relapse may be still considered for a salvage concurrent chemo-radiation approach

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Chiappori, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination Immunotherapy Plus Vaccine
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Combination Immunotherapy Plus Vaccine
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR)
Description: Response will be assessed primarily using the response evaluation criteria in solid tumors (RECIST v1.1). The immune related (ir)RECIST will also be used secondarily. DCR = Complete Response (CR) = Partial Response (PR) + Stable Disease (SD) rates. The disease control (DCR=CR+PR+SD) rates will be summarized using both point estimates and exact confidence intervals based on the binomial distribution by group.
Time Frame: Up to 3 years
Population: Evaluable participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Immunotherapy Plus Vaccine
Number analyzed (Participants) | 11
percentage of participants | 42.85 [21.3 to 67.4]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: The PFS, defined as time from enrollment (eligible date) to date of progression/death, whichever happens first, or censor at last clinical follow-up date. PFS will be summarized utilizing the K-M method.
Time Frame: Up to 3 years
Population: Evaluable participants
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Combination Immunotherapy Plus Vaccine
Number analyzed (Participants) | 14
days | 63 [56 to 334]

3. Secondary Outcome: Overall Survival (OS)
Description: The OS, defined as the time from study enrollment (eligible date) to death from any cause. OS will be summarized utilizing the K-M method.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Combination Immunotherapy Plus Vaccine
Number analyzed (Participants) | 14
days | 120 [67 to NA] — upper limit was not reached

4. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR=CR+PR) will be summarized using both point estimates and exact confidence intervals based on the binomial distribution by group.
Time Frame: Up to 3 years
Population: Evaluable participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Immunotherapy Plus Vaccine
Number analyzed (Participants) | 11
percentage of participants | 21.4 [7.57 to 47.5]

ADVERSE EVENTS:
Time Frame: Adverse Events collected from date of participant consent to 30 days post last treatment. (an average of 1 year). Survival was assessed up to 3 years.
Arm/Group | Combination Immunotherapy Plus Vaccine
All-Cause Mortality (participants affected / at risk) | 12/14
Serious Adverse Events (participants affected / at risk) | 14/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Immunotherapy Plus Vaccine (N=14)
Platelet count decreased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) — Diabetic ketoacidosis
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Investigations - Other (Investigations) | 1 (1) — Pancytopenia
Death NOS (General disorders) | 3 (3)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (2)
Psychiatric disorders -Other (Psychiatric disorders) | 1 (1) — Altered mental status
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1) — Cholecystitis
Infections and Infestations - Other (Infections and infestations) | 1 (1) — Enteritis
Renal and urinary disorders -Other (Renal and urinary disorders) | 1 (1) — Medical renal disease
Seizure (Nervous system disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) — Death due to disease progression
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Immunotherapy Plus Vaccine (N=14)
Fatigue (General disorders) | 8 (8)
Pain (General disorders) | 6 (9)
Chills (General disorders) | 3 (3)
Fever (General disorders) | 2 (2)
Edema face (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (12)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 5 (12)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (5)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (5)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 2 (2)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 4 (8)
Constipation (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (7)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (7)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 5 (9)
Weight loss (Investigations) | 4 (10)
Alanine aminotransferase increased (Investigations) | 3 (10)
Aspartate aminotransferase increased (Investigations) | 3 (11)
Blood bilirubin increased (Investigations) | 2 (3)
Lipase increased (Investigations) | 2 (3)
Cholesterol high (Investigations) | 1 (2)
Creatinine increased (Investigations) | 1 (1)
Investigations - Other (Investigations) | 1 (2)
Lymphocyte count decreased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 1 (2)
Serum amylase increased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 5 (5)
Dysgeusia (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 2 (3)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (8)
Leukocytosis (Blood and lymphatic system disorders) | 2 (3)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Cardiac disorders - Other (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Confusion (Psychiatric disorders) | 3 (5)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Infections and infestations - Other (Infections and infestations) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (3)
Hematuria (Renal and urinary disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/15/NCT03406715/Prot_SAP_000.pdf